CLINICAL TRIAL: NCT06587594
Title: Supportive Outcomes Through Listening, Validation, and Empowerment
Acronym: SOLVE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Sandy Magaña, Professor, University of Texas at Austin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00006256
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-07

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: autism, mental health, solution focused brief therapy, autistic adults
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder; Psychological Well-Being | interventions — Psychotherapy, Brief

STUDY DESIGN:
Intervention Model Description: One group pre and post-test design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SFBT intervention (Experimental): Behavioral: Solution-focused Brief Therapy (SFBT) A behavioral health intervention designed to help autistic adults to make a positive change in their life using strength-based approach.
  Interventions: Behavioral: Solution Focused Brief Therapy

INTERVENTIONS:
Behavioral: Solution Focused Brief Therapy — A behavioral health intervention designed to help autistic adults to make a positive change in their life using strength-based approach.

SUMMARY:
This research aims to pilot an intervention that will provide practitioners and clinicians with evidenced-based behavioral health strategies for working with autistic adults. The findings will contribute to the needed, yet sparse research of evidence-based behavioral health interventions for this population.

The guiding research aims for this study are:

1. To implement a small-scale pilot study aimed at refining the Solution Focused Brief Therapy (SFBT) and protocol for use with autistic adults based on clinician expertise and lived experience.
2. To test the feasibility and acceptability of the SFBT. Namely, how well the intervention is received by this population and if participants can attend and engage in all 4 sessions.
3. To evaluate outcomes before and after the intervention and assess for any improvements through valid and reliable measurements of behavioral health outcomes.

This research aims to answer the following research questions:

1. What is the retention rate of participants in the 4-weekly sessions of the SOLVE program?
2. Do participants show progress in their self-identified goals after the intervention?
3. What are the experiences and satisfaction rates of participants in participating in a four-session SFBT intervention?
4. Do participants report higher scores in quality of life and lower depressive and anxiety scores between baseline and immediately post-intervention?

The five autistic participants will participate in four one-on-one weekly SFBT sessions conducted by licensed mental health professionals. The intervention is expected to take four to 5 weeks, allowing for cancelations and rescheduling as needed.

DETAILED DESCRIPTION:
Step 1 of the first SFBT session: Introduction to SFBT Sessions and Agenda-setting The first SFBT session will include the introduction to SFBT sessions and agenda setting. The SFBT session and agenda description can be written down and given to the participants to read, take home, or be provided ahead of time in writing. The participants will be given time to ask questions.

Step 2 of the first SFBT session: Exploration of Strengths, Interests, and Support Systems After introducing the SFBT sessions, the clinician will ask about the participant's strengths, interests, and support systems. The goal of this phase should be to identify participant strengths, interests, and support systems. The participants will be reassured that they can take their time and that there are no right or wrong answers. The participants will be offered the option to use their preferred method of response and communication. The clinician will document the participant's chosen method of response and communication to maintain consistency and track preferences. The participant will be given the option to choose from multiple choice options if they are finding it challenging to answer the open-ended questions. The multiple-choice options will include an open-ended response.

Step 3 of the first SFBT session: Goal Exploration and Definition The clinician will invite the participant to develop a session topic and state their goal for the meeting. The goal will come from the participant and be co-constructed with the clinician. The goal will be described in concrete and behavioral terms. If the participant is finding it challenging to answer these open-ended, the clinician may offer multiple choice as examples or options but will be careful to not direct the participant.

Step 4 of the first SFBT session: Description of a Preferred Future The participant will describe in detail what their life will be like when they have reached their goal. The clinician will use concrete language defining each word. During the session the clinician will use a daily log to ask the participant to describe what they are doing differently at time points in the day.

Step 5 of the first SFBT session: Exploring Exceptions The clinician will help the participants identify exceptions to the problem or times when the problem has been less noticeable or is a little better for them.

Step 6 of the first SFBT session: Scaling Questions The clinicians ask the participants scaling questions to help the participants to anchor their problems or goals with descriptions on a scale and to use that rating to ask them what it will take for them to move forward to the next step. The participants will be offered to use a visual scale with pictures to represent the numbers.

Study Design. The study uses a one group pretest posttest design to assess and evaluate the feasibility and acceptability of Solution-Focused Brief Therapy (SFBT) in autistic adults. We will utilize both quantitative and qualitative measures to assess baseline and outcome. The study aims to recruit five autistic adults to participate in the pilot SFBT sessions in collaboration with community organization. Participants will undergo virtual screening (on the UT Zoom platform) and in-person pre-assessments before the first SFBT session. The assessments and four SFBT sessions will be conducted in-person. Each participant will undergo four in-person one-on-one SFBT sessions conducted by licensed mental health professionals. Post-assessments will be conducted in-person after the last SFBT session.

Data Analysis. Our main aims are to assess feasibility and acceptability. Feasibility will be determined by the number of eligible participants recruited to the study, the number of participants who completed all four sessions, and for those who didn't the number of sessions completed. Retention rates will be calculated by dividing the number that completed 4 sessions by 4.

Acceptability will be assessed using the open-ended questions in the interviews. To analyze open-ended questions, we will use a mixed approach combining inductive reasoning with predetermined codes related to the acceptability and satisfaction of the intervention (Tariq & Woodman, 2013).

Secondary aims are to determine whether there are changes between pre and post-test that show promising trends.

All demographic variables (e.g. race/ethnicity, sex, sexual orientation, employment status, education level) will be summarized by standard descriptive statistics (means and standard deviations for continuous variables and frequencies for categorial variables). As the sample size is small, inferential analyses will be approached with caution. Assumptions for parametric analyses will be checked; if violated, nonparametric methods will be considered.

We will calculate summary statistics for total scores and scores on individual items on outcome measures. We will assess the normality of the differences between the pre and post test scores. We will analyze the pre and post scores using either a paired-sample t-test or the Wilcoxon signed-rank test depending on the distributional characteristics of the data. Effect sizes will be calculated.

Study measures. Social Responsiveness Scale Short Form (16 items): This scale is used with autistic individuals to identify and quantify the severity of social impairment. A study on a large sample of youth from four ASD databases demonstrated that the Social Responsiveness Scale Short Form (SRS-SF) has high reliability, with a Cronbach's alpha coefficient of 0.96, indicating strong internal consistency. The study suggested validity with the SRS-SF showing strong relationships with established measures of ASD severity, including the Autism Diagnostic Observation Schedule (ADOS), Autism Diagnostic Interview-Revised (ADI-R), and Vineland Adaptive Behavior Scales. This suggests that the SRS-SF effectively captured core symptoms of ASD (Sturm et al., 2017).

Demographics and Household SES: A study-specific demographics questionnaire will be developed to capture background information. The demographic questions will take participants approximately 10 minutes to complete and will include sex and gender identity, SES, race/ethnicity, co-morbid ADHD and mental health diagnoses. Anxiety Scale for Adults-Autism The Anxiety Scale for Adults- Autism is a 20 item self-reported measure consisting of a General Anxiety Factor and three group factors: Social Anxiety, Anxious Arousal, and Uncertainty (Rodgers et al).

Depression Scale for Adults-Autism (ADAT-A): The ADAT-A is a self-reported 21 items measure designed with feedback from autistic adults, based on DSM-V and ICD-10 criteria for depression and adapted from the PHQ9. There are three subscales: Cognitive/Affective symptoms of depression according to DSM-V/ICD-10 criteria, Somatic symptoms of depression according to DSM-V/ICD-10 criteria and Autistic, autism-specific signs of depression (Cassidy et al).

PROMIS General Life Satisfaction- Short Form: The PROMIS General Life Satisfaction Short Form questionnaire is a 4 item self-reported measure assessing how much one agrees with each item in general rather than over a specified time period (PROMIS).

PROMIS Positive Affect Short Form: The PROMIS Positive Affect Short Form is a 15 item self-reported measure that assesses positive emotional experiences.

Open-ended questions: Before the SBFT sessions, we will ask participants questions regarding their current concerns, strengths and resources, expectations and goals, session feedback, and future outlook. After completing the four sessions, we will ask similar questions to see if there are any behavioral changes.

Post-intervention open ended questions:

1. Current Concerns - Reflecting on the past sessions, have there been any changes in the challenges or difficulties you mentioned at the beginning?
2. Strengths and Resources - Have you noticed any new strengths or resources that you did not recognize before starting the sessions?
3. Expectations and Goals - Looking back, have your expectations or goals for the therapy been met? If so, how?
4. Session Feedback - How would you describe your overall experience during the therapy sessions? What aspects did you find helpful or challenging? How do you feel about the number of SFBT sessions you received? What do you want to improve?
5. Future Outlook - After completing the therapy sessions, how do you see yourself moving forward? What changes, if any, do you anticipate?

ELIGIBILITY:
Inclusion Criteria:

1. Autism diagnosis by a medical, mental health, or school professional
2. Between the ages of 18 and 30 years old
3. Proficient in English
4. Able to communicate verbally
5. Able to attend assessment and therapy sessions in person in a Center in Austin
6. Willing to complete two assessment sessions and 4 in-person therapy sessions

Exclusion Criteria:

* screen positive for suicidal ideation
* currently being treated for major mental health condition (medication or behavior intervention)
* has a legal guardian designated by the court

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
PROMIS General Life Satisfaction | Change from baseline positive affect at one month
  minimum 4 maximum 9, higher scores indicate higher general life satisfaction
PROMIS Positive Affect - Short Form | Change from baseline positive affect at one month
  minimum 15 maximum 75; higher scores indicate higher positive affect

SECONDARY OUTCOMES:
Anxiety Scale for Adults - Autism | Change from baseline depression at one month
  minimum 20 maximum 80, higher scores indicate greater levels of anxiety
Depression Scale for Adults - Autism | Change from baseline depression at one month
  minimum 21 maximum 84, higher scores indicate greater levels of depression

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas, Texas Center for Disability Studies, Austin, Texas, United States

IPD SHARING:
Plan to Share IPD: No
This is a small pilot study